CLINICAL TRIAL: NCT01051557
Title: Phase I/II Trial of Temsirolimus and Perifosine for Recurrent or Progressive Malignant Gliomas
Brief Title: Temsirolimus and Perifosine in Treating Patients With Recurrent or Progressive Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01409; NCI-2011-01409 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-058; MSKCC-09058; CDR0000663573; 09-058 (Other: Memorial Sloan Kettering Cancer Center); 8249 (Other: CTEP); P30CA008748 (NIH); U01CA069856 (NIH)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Diffuse Astrocytoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Adult Oligodendroglioma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — perifosine; octadecyl-(N,N-dimethylpiperidino-4-yl)-phosphate; temsirolimus; Sirolimus

ARMS (1):
- Treatment (temsirolimus and perifosine) (Experimental): PHASE I: Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22 and perifosine PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients receive temsirolimus and perifosine as in phase I. Some patients may also undergo cytoreductive surgery.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Perifosine; Drug: Temsirolimus; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Perifosine — Given PO
  Other Names: 4-[[Hydroxy(octadecyloxy)phosphinyl]oxy]-1,1-dimethylpiperidinium, Inner Salt; D21266; Octadecylphosphopiperidine
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
Procedure: Therapeutic Conventional Surgery — Undergo cytoreductive surgery

SUMMARY:
This phase I/II trial studies the side effects and best dose of temsirolimus when given together with perifosine and to see how well it works in treating patients with recurrent or progressive malignant glioma. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as perifosine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving temsirolimus with perifosine may be an effective treatment for malignant glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Define the maximum tolerated dose (MTD) of temsirolimus in combination with perifosine in patients with recurrent or progressive malignant glioma who are not taking enzyme-inducing anti-epileptic drugs (EIAEDs). (Phase I) II. Determine the efficacy of temsirolimus in combination with perifosine in patients with recurrent/progressive glioblastomas (GBMs) not taking EIAEDs as measured by 6 month progression-free survival (6mPFS) and radiographic response rates. (Phase II)

SECONDARY OBJECTIVES:

I. Characterize the safety profile of perifosine and temsirolimus. II. Estimate median overall and progression-free survival. III. Explore the association of pre-treatment molecular phenotype with response to treatment.

IV. Explore molecular effects during treatment including phosphatidylinositol-3 kinase (PI3K)/protein kinase B (AKT)/mammalian target of rapamycin (mTOR)/ribosomal protein S6 kinase (S6K) and rat sarcoma (RAS)/mitogen-activated protein kinase kinase (MEK)/mitogen-activated protein kinase (ERK) signaling, proliferation, and apoptosis.

OUTLINE: This is a phase I dose-escalation study of temsirolimus, followed by a phase II study.

PHASE I: Patients receive temsirolimus intravenously (IV) over 30 minutes on days 1, 8, 15, and 22 and perifosine orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients receive temsirolimus and perifosine as in phase I. Some patients may also undergo cytoreductive surgery.

After completion of study therapy, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have unstained slides or tissue blocks available from at least one prior surgery; frozen tissue is also requested if available
* Patients must have received prior radiotherapy and temozolomide; there is otherwise no limit on the number of prior recurrences/therapies
* At least 6 weeks (42 days) must have elapsed since completion of radiation therapy to initiation of study treatment
* At least 4 weeks (28 days) must have elapsed since most recent temozolomide and initiation of study treatment
* Patients must have recovered from the toxic effects of other prior direct inhibitors of vascular endothelial growth factor (VEGF)/VEGF receptor (VEGFR): 4 weeks from prior therapy with agents such as bevacizumab (Avastin), aflibercept (VEGF-Trap), cediranib (AZD2171), or XL-184 (BMS 907351); any questions regarding the definition of a direct anti-VEGF/VEGFR therapy must be discussed with the principal investigator (PI) or co-PI; patients must have recovered from the toxic effects of other prior therapy including: 4 weeks (28 days) from any investigational agent, two weeks (14 days) from vincristine, 6 weeks (42 days) from nitrosoureas, 3 weeks (21 days) from procarbazine administration, and 1 week (7 days) for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count), and 4 weeks (28 days) from any other prior cytotoxic therapy; any questions related to the definition of non-cytotoxic agents should be directed to the co-PI
* Patients must have shown unequivocal evidence for tumor progression by magnetic resonance imaging (MRI)/computed tomography (CT) on the baseline MRI/CT in comparison to a prior scan OR have recently undergone resection for recurrent/progressive disease; the baseline brain MRI/CT must be performed 14 days or fewer prior to treatment; the same type of scan, i.e., MRI (or CT for patients who cannot undergo MRI) must be used throughout the period of protocol treatment for tumor measurement; criteria for progression on this study are not mandatory if the disease progression is obvious in the opinion of the investigator; any questions should be addressed to the PI
* Patients must be on a stable or decreasing dose of corticosteroids for a minimum of 5 days before the baseline MRI/CT (and positron emission tomography [PET] scans for patients on the phase II study) except patients undergoing surgery on the surgical substudy of phase II; if the corticosteroid dose is increased between the date of imaging and registration a new baseline MR/CT is required
* Karnofsky performance status >= 60%
* Life expectancy of greater than 8 weeks
* White blood cell (WBC) >= 2,000/ul
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count of >= 100,000/mm^3

  * Platelet count of at least 100,000/mm^3 on at least 2 consecutive blood draws, at least 1 week apart, with results stable/trending upward; any question regarding the definition of stable/trending upward must be discussed with the PI
* Hemoglobin >= 10 gm/dl; eligibility level for hemoglobin may be reached by transfusion
* Serum glutamic oxaloacetic transaminase (SGOT), serum glutamate pyruvate transaminase (SGPT) < 2 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* Creatinine < 1.5 mg/dL
* Calcium levels at or above the lower limit of normal
* Phosphorus levels at or above the lower limit of normal
* Cholesterol level =< 350 mg/dl
* Triglycerides level =< 400 mg/dl
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Women of childbearing potential must have a negative beta-human chorionic gonadotropin (B-HCG) pregnancy test documented within 7 days prior to treatment
* Women must agree not to breast feed
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Measurable disease is not required for eligibility in patients who recently underwent resection as long as progressive disease led to the surgery, and the histology of the most recent surgery documented recurrent/progressive/persistent malignant glioma

  * If cytoreductive surgery is planned for tumor recurrence at the time of enrollment, such patients may be eligible for the surgical substudy (Phase II only), taking temsirolimus + perifosine pre-operatively and then re-initiating such therapy after recovering from the effects of surgery
* PHASE I: Patients must have a EITHER

  * Histologically confirmed intracranial malignant glioma of the following types: glioblastoma, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic oligo-astrocytoma (AOA) also called anaplastic mixed gliomas, malignant glioma NOS (not otherwise specified); patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a high grade (malignant) glioma is made; OR
  * Histologically confirmed low grade (World Health Organization [WHO] grade II) gliomas (such as low grade astrocytoma, low grade oligodendroglioma, low grade oligo-astrocytoma (mixed gliomas), or low grade glioma NOS) IF there is radiographic evidence by MRI or CT of malignant transformation but histologic confirmation of high grade (malignant) transformation would not be otherwise undertaken for routine clinical care; inclusion of patients in this group will allow increased accrual rapidity by enrolling patients who are otherwise ineligible for almost all malignant glioma trials yet whom are treated presumptively for malignant glioma
* PHASE II: Patients must have a histologically confirmed intracranial malignant glioma of the following types: glioblastoma, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic oligo-astrocytoma (AOA) also called anaplastic mixed gliomas, malignant glioma NOS (not otherwise specified); patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a high grade (malignant) glioma is made
* PHASE II (patients enrolling on the surgical substudy to evaluate tissue correlates): Patients eligible for the surgical subset have been identified as candidates for cytoreductive surgery by the treating physician and/or based on discussion in a multidisciplinary tumor board, with the input of other surgeons as well as that of the neuro-oncologists involved in the trial; for the patients in the preoperative component, a scan showing progression is required but stable corticosteroids are not required; following surgery, a scan should be done less than 96 hours after surgery; if this is not performed, then a new baseline scan should be performed at least 4 weeks after surgery to avoid misinterpretation of post-operative changes as enhancing disease; this scan will serve as the new baseline before restarting treatment post-operative, and it must be performed on a stable or decreasing dose of corticosteroids; (as above, regarding the baseline MRI or CT scan prior to registration, patients in the Phase II component who are NOT participating in the pre-operative component of the study should be on a steroid dose that has been stable for at least 5 days prior to the scan; if the corticosteroid dose is increased between the date of imaging and registration a new baseline MR/CT is required)
* PHASE II (patients enrolling on the surgical substudy to evaluate tissue correlates): Post-operatively, treatment with temsirolimus and perifosine must re-start no later than the 14th day after the scan; if the 96-hour scan is more than 14 days old before treatment is initiated, the scan needs to be repeated on a stable or decreasing steroid dose; treatment must start no later than 56 days after surgery
* PHASE II (patients previously treated with bevacizumab or other direct inhibitors of VEGF/VEGFR including Aflibercept (VEGF-Trap) and cediranib and XL-184 (BMS 907351): There is no limit on such therapy for patients accrued to phase I; for phase II, historical controls for this group of patients is poorly defined; therefore, we will accrue up to 15 patients who received prior treatment with direct VEGF/VEGFR inhibitors in order to gain preliminary data for use as a comparison group in a follow up study; all other inclusion/exclusion criteria also apply to this cohort

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to temsirolimus or perifosine
* Patients must not be taking EIAED; if previously on an EIAED, the patient must be off of it for at least two weeks prior to treatment on study
* Patients must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with temsirolimus and perifosine
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* PHASE II: Patients may not have received prior treatment with mTOR inhibitors such as temsirolimus, rapamycin (sirolimus), or RAD001 (everolimus); any question regarding the definition of mTOR inhibiting therapy must be discussed with the PI; such prior therapy is allowed for the phase I component
* PHASE II: Patients may not have previously received perifosine or other AKT targeting agents; any question regarding the definition of AKT targeting therapy must be discussed with the PI; such prior therapy is allowed for the phase I component
* PHASE II: Patients must not have received prior treatment with convection enhanced delivery, other catheter based intra-tumoral treatment, or carmustine (BCNU)/Gliadel wafers; such prior therapy is allowed for the phase I component
* PHASE II: Patients with prior therapy that included stereotactic radiosurgery (including gamma-knife or cyber-knife) during therapy for newly diagnosed or recurrent disease, or re-irradiation of any type, must have confirmation of true progressive disease rather than radiation necrosis based upon surgical documentation of recurrent/progressive disease; imaging with magnetic resonance (MR) spectroscopy, PET, or other techniques is not adequate to exclude radiation necrosis for this study; such prior therapy is allowed for the phase I component and does not require surgical documentation of disease
* PHASE II: Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible for the phase II study but are eligible for the phase I component

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-01-27 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Kaley, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 (Temsirolimus: 15 mg/wk): Cycle = 28 days: Cycle 1 Temsirolimus: 15 mg/wk IV over 30 min Perifosine: 600 mg loading dose PO on day 1and maintence dose 100 mg PO QD on days 2-28, Cycle 2+ Temsirolimus: 15 mg/wk IV over 30 min Perifosine: 100 mg maint dose PO QD on days 1-28
- 2 (Temsirolimus: 25 mg/wk): Cycle = 28 days: Cycle 1 Temsirolimus: 25 mg/wk IV over 30 min Perifosine: 600 mg loading dose PO on day 1and maintence dose 100 mg PO QD on days 2-28, Cycle 2+ Temsirolimus: 25 mg/wk IV over 30 min Perifosine: 100 mg maint dose PO QD on days 1-28
- 3 (Temsirolimus: 50 mg/wk): Cycle = 28 days: Cycle 1 Temsirolimus: 50 mg/wk IV over 30 min Perifosine: 600 mg loading dose PO on day 1and maintence dose 100 mg PO QD on days 2-28 Cycle 2+ Temsirolimus: 50 mg/wk IV over 30 min Perifosine: 100 mg maint dose PO QD on days 1-28
- 4 (Temsirolimus: 75 mg/wk): Cycle = 28 days: Cycle 1 Temsirolimus: 75 mg/wk IV over 30 min Perifosine: 600 mg loading dose PO on day 1and maintence dose 100 mg PO QD on days 2-28, Cycle 2+ Temsirolimus: 75 mg/wk IV over 30 min Perifosine: 100 mg maint dose PO QD on days 1-28
- 5 (Temsirolimus: 115 mg/wk): Cycle = 28 days: Cycle 1 Temsirolimus: 115 mg/wk IV over 30 min Perifosine: 600 mg loading dose PO on day 1and maintence dose 100 mg PO QD on days 2-28, Cycle 2+ Temsirolimus: 115 mg/wk IV over 30 min Perifosine: 100 mg maint dose PO QD on days 1-28
- 6 (Temsirolimus: 170 mg/wk): Cycle = 28 days: Cycle 1 Temsirolimus: 170 mg/wk IV over 30 min Perifosine: 600 mg loading dose PO on day 1and maintence dose 100 mg PO QD on days 2-28, Cycle 2+ Temsirolimus: 170 mg/wk IV over 30 min Perifosine: 100 mg maint dose PO QD on days 1-28
- 7 (Temsirolimus: 170 mg/wk Perifosine: 900 mg Loading Dose ): Cycle = 28 days: Cycle 1 Temsirolimus: 170 mg/wk IV over 30 min Perifosine: 900 mg loading dose PO on day 1and maintence dose 100 mg PO QD on days 2-28 Cycle 2+ Temsirolimus: 170 mg/wk IV over 30 min Perifosine: 100 mg maint dose PO QD on days 1-28
Period: Overall Study
Arm/Group | 1 (Temsirolimus: 15 mg/wk) | 2 (Temsirolimus: 25 mg/wk) | 3 (Temsirolimus: 50 mg/wk) | 4 (Temsirolimus: 75 mg/wk) | 5 (Temsirolimus: 115 mg/wk) | 6 (Temsirolimus: 170 mg/wk) | 7 (Temsirolimus: 170 mg/wk Perifosine: 900 mg Loading Dose )
Started | 4 | 3 | 6 | 3 | 8 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 4 | 3 | 6 | 3 | 7 | 6 | 6
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — disease progression | 3 | 3 | 5 | 2 | 4 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 (Temsirolimus: 15 mg/wk) | 2 (Temsirolimus: 25 mg/wk) | 3 (Temsirolimus: 50 mg/wk) | 4 (Temsirolimus: 75 mg/wk) | 5 (Temsirolimus: 115 mg/wk) | 6 (Temsirolimus: 170 mg/wk) | 7 (Temsirolimus: 170 mg/wk Perifosine: 900 mg Loading Dose ) | Total
Number analyzed (Participants) | 4 | 3 | 6 | 3 | 8 | 6 | 6 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6 | 3 | 7 | 5 | 5 | 32
  >=65 years | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 2 | 3 | 2 | 0 | 12
  Male | 3 | 2 | 3 | 1 | 5 | 4 | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 4 | 3 | 6 | 2 | 6 | 6 | 6 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 5 | 3 | 7 | 6 | 5 | 31
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 6 | 3 | 8 | 6 | 6 | 36

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Temsirolimus
Description: MTD defined as the dose at which fewer than one-third of patients experience a dose limiting toxicity (DLT) according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (Phase I)
Time Frame: 28 days
Measure: Number; unit: mg/week
Arm/Group | Treatment (Temsirolimus and Perifosine)
Number analyzed (Participants) | 36
mg/week | 115

2. Primary Outcome: Determine the Efficacy of Temsirolimus in Combination With Perifosine in Patients With Recurrent/Progressive Glioblastomas (GBMs) Not Taking EIAEDs as Measured by 6 Month Progression-free Survival (6mPFS) and Radiographic Response Rates. (Phase II)
Time Frame: 5 years
Population: Data were not collect as as study did not progress to Phase II.
Arm/Group | 1 (Temsirolimus: 15 mg/wk) | 2 (Temsirolimus: 25 mg/wk) | 3 (Temsirolimus: 50 mg/wk) | 4 (Temsirolimus: 75 mg/wk) | 5 (Temsirolimus: 115 mg/wk) | 6 (Temsirolimus: 170 mg/wk) | 7 (Temsirolimus: 170 mg/wk Perifosine: 900 mg Loading Dose )
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | 1 (Temsirolimus: 15 mg/wk) | 2 (Temsirolimus: 25 mg/wk) | 3 (Temsirolimus: 50 mg/wk) | 4 (Temsirolimus: 75 mg/wk) | 5 (Temsirolimus: 115 mg/wk) | 6 (Temsirolimus: 170 mg/wk) | 7 (Temsirolimus: 170 mg/wk Perifosine: 900 mg Loading Dose )
All-Cause Mortality (participants affected / at risk) | 4/4 | 3/3 | 6/6 | 2/3 | 7/8 | 6/6 | 6/6
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 1/6 | 1/3 | 3/8 | 4/6 | 3/6
Other Adverse Events (participants affected / at risk) | 4/4 | 2/3 | 6/6 | 3/3 | 7/8 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 (Temsirolimus: 15 mg/wk) (N=4) | 2 (Temsirolimus: 25 mg/wk) (N=3) | 3 (Temsirolimus: 50 mg/wk) (N=6) | 4 (Temsirolimus: 75 mg/wk) (N=3) | 5 (Temsirolimus: 115 mg/wk) (N=8) | 6 (Temsirolimus: 170 mg/wk) (N=6) | 7 (Temsirolimus: 170 mg/wk Perifosine: 900 mg Loading Dose ) (N=6)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 (Temsirolimus: 15 mg/wk) (N=4) | 2 (Temsirolimus: 25 mg/wk) (N=3) | 3 (Temsirolimus: 50 mg/wk) (N=6) | 4 (Temsirolimus: 75 mg/wk) (N=3) | 5 (Temsirolimus: 115 mg/wk) (N=8) | 6 (Temsirolimus: 170 mg/wk) (N=6) | 7 (Temsirolimus: 170 mg/wk Perifosine: 900 mg Loading Dose ) (N=6)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Cholesterol high (Investigations) | 1 (3) | 2 (6) | 1 (2) | 2 (8) | 2 (13) | 3 (6) | 3 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (2) | 1 (5) | 4 (6) | 3 (4) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 4 (9) | 3 (4) | 3 (5) | 4 (6) | 1 (7)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 3 (19) | 1 (1) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 3 (12) | 2 (4) | 2 (12)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (15) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (5) | 2 (7)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 3 (8) | 1 (2) | 3 (5) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 1 (2)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ejaculation disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT01051557/Prot_SAP_000.pdf